CLINICAL TRIAL: NCT02934633
Title: Parent Training in Child Safety Practices
Acronym: BabySafety_2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Center for Applied Science, Inc. (Industry)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: SBIR 63-2; R44HD044281 (NIH)
Record Dates: First submitted 2013-05-31; First posted 2016-10-17 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Injury
Keywords: injury; child; cars; pedestrians; child safety; interactive; computer; prevention; internet; CD-ROM
MeSH Terms: conditions — Wounds and Injuries | interventions — tyrosyl-1,2,3,4-tetrahydro-3-isoquinolinecarbonyl-phenylalanyl-phenylalanine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Keeping Baby Safe (Experimental): Keeping Baby Safe 2-DVD package, designed for parents of children from birth to 24 months. One DVD addresses automobile passenger safety and focuses on the correct choice and proper installation of child safety seat for the age of the parent's child. The second DVD covers a core set of home safety skills: (a) preventing falls, (b) preventing fires and burns, (c) preventing poisoning, (d) firearm safety, (e) preventing drowning, (f) preventing suffocation and choking, (e) play equipment safety, and (f) animal safety. Content in the home safety DVD is based on information the American Academy of Pediatrics (AAP) recommends that physicians provide to parents during well-baby visits.
  Interventions: Behavioral: Keeping Baby Safe 2-DVD package
- AAP TIPP Sheets (Active Comparator): American Academy of Pediatrics The Injury Prevention Program (TIPP) sheets. Paper-based information sheets that parents would typically receive from their pediatrician or general practitioner at well-baby visits.
  Interventions: Behavioral: The Injury Prevention Program (TIPP) sheets

INTERVENTIONS:
Behavioral: Keeping Baby Safe 2-DVD package — Keeping Baby Safe is a 2-DVD package that teaches childhood injury prevention skills to parents of children from birth to 24 months of age. One DVD addresses automobile passenger safety and focuses on the correct choice and proper installation of child safety seat for the age of the parent's child. The second DVD covers a core set of home safety skills: (a) preventing falls, (b) preventing fires and burns, (c) preventing poisoning, (d) firearm safety, (e) preventing drowning, (f) preventing suffocation and choking, (e) play equipment safety, and (f) animal safety. Content in the home safety DVD is based on information the American Academy of Pediatrics (AAP) recommends that physicians provide to parents during well-baby visits.
  Arms: Keeping Baby Safe
Behavioral: The Injury Prevention Program (TIPP) sheets — American Academy of Pediatrics The Injury Prevention Program (TIPP) sheets. Paper-based information sheets parents would typically receive from their pediatrician or general practitioner at well-baby visits.
  Arms: AAP TIPP Sheets

SUMMARY:
This project completed an intervention designed to teach parents of children aged 0-2 years of age how to prevent injuries to their child. The intervention consisted of a two DVD package with information on creating a safe home environment and correctly choosing and installing an appropriate car safety seat. The study hypothesis was that parents who used the intervention would score significantly higher on measures of knowledge, motivation, intention and self-efficacy in implementing injury prevention strategies.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Parent whose oldest child is 0-24 months old
* Speak and read English
* Have internet access (online study only)

Exclusion Criteria:

* Parents who do not have legal or physical custody
* Subjects live in a household in which a family member had an overnight stay in the hospital as a result of an injury in the last 2 years

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 414 (Actual)
Dates: Start 2006-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Change in parent motivation to implement injury prevention strategies | 7 day and 30 day post intervention
Change in parent knowledge of injury prevention practices | 7 and 30 day post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lynne H Grilley Swartz, MPH, CHES, Principal Investigator — Oregon Center for Applied Science
Locations (1):
- Oregon Center for Applied Science, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No